CLINICAL TRIAL: NCT01573676
Title: The Influence of Bariatric Surgery on Patients With Obstructive Sleep Apnea (OSA)
Acronym: OSA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0048-11-HYMC
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-04

CONDITIONS: Overweight; Obstructive Sleep Apnea
Keywords: bariatric surgery; sleep apnea; overweight
MeSH Terms: conditions — Overweight; Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bariatric surgery patients: Candidates for bariatric surgery.

SUMMARY:
Obesity is a very important risk-factor in obstructive sleep apnea (OSA) and other sleep breathing disorders in patients with extreme BMI.

Candidates for bariatric surgery have a high OSA prevalence, ranging from 60-83%. The characteristics of patients with sleep apnea that were evaluated for bariatric surgery and had a full overnight polysomnography (PSG) screening for OSA were described and it was found that a very high prevalence (77.2%) for OSA in all subjects evaluated, regardless of pre-operative risk for OSA. A post-bariatric surgery PSG was not a part of this study.

The investigators would like to demonstrate the impact of bariatric surgery on OSA as a function of time.

ELIGIBILITY:
Inclusion Criteria:

* All candidates for bariatric surgery over 18 yrs of age

Exclusion Criteria:

* Patients that underwent any OSA surgery in the past
* Patient had any bariatric surgery in the past
* Patients with COPD
* Patients with CHD
* Patients who have / had cancer that received chemotherapy or radiotherapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: both males and females
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in RDI after bariatric surgery | Six months
  Improvement will measured by polysonography